CLINICAL TRIAL: NCT01326780
Title: A Multi-Center, Double-Blind, Vehicle Controlled, Phase II Study of JNJ 10229570-AAA for the Treatment of Acne Vulgaris
Brief Title: A Study of a New Drug Treatment for Acne
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA-P-8023
Record Dates: First submitted 2011-03-30; First posted 2011-03-31 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Acne Vulgaris
Keywords: Acne; Irritation; Safety; Sebum
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1.2% Facial Cream (Experimental): 1.2% JNJ 10229570-AAA
  Interventions: Drug: 1.2% JNJ 10229570-AAA
- 2.4% Facial Cream (Experimental): 2.4% JNJ 10229570-AAA
  Interventions: Drug: 2.4% JNJ 10229570-AAA
- 3.6% Facial Cream (Experimental): 3.6% JNJ 10229570-AAA
  Interventions: Drug: 3.6% JNJ 10229570-AAA
- 0% Facial Cream (Placebo Comparator): Vehicle control
  Interventions: Other: Vehicle control

INTERVENTIONS:
Drug: 1.2% JNJ 10229570-AAA — 1.2% JNJ 10229570-AAA 1.2% cream applied once daily to the face for 12 weeks
  Other Names: Not yet marketed
  Arms: 1.2% Facial Cream
Drug: 2.4% JNJ 10229570-AAA — 2.4% JNJ 10229570-AAA 2.4% cream applied once daily to the face for 12 weeks
  Other Names: Not yet marketed
  Arms: 2.4% Facial Cream
Drug: 3.6% JNJ 10229570-AAA — 3.6% JNJ 10229570-AAA 3.6% cream applied once daily to the face for 12 weeks
  Other Names: Not yet marketed
  Arms: 3.6% Facial Cream
Other: Vehicle control — Color matched cream vehicle, applied once daily to the face for 12 weeks
  Other Names: Not marketed
  Arms: 0% Facial Cream

SUMMARY:
A study to determine if three different doses of a new acne treatment are safe and better at reducing facial acne than a treatment without active ingredient.

DETAILED DESCRIPTION:
Approximately 400 male and female subjects with moderate facial acne vulgaris will be enrolled in this randomized, multi-center study. Following satisfaction of entry criteria and screening procedures, subjects will be randomized to either 1.2%, 2.4%, or 3.6% facial cream (JNJ 10229570-AAA) or color-matched vehicle. Subjects will apply the study medication once daily on the face for 12 weeks. Safety will be monitored throughout the study duration. Efficacy will be assessed by facial lesion counts and by the investigator global evaluation of acne severity at Baseline and at Weeks 2, 4, 6, 8, 10, and 12. Approximately 50 subjects from one investigational site also will have serums collected at Weeks 6 and 12 for evaluation of the multiple dose pharmacokinetics of JNJ 10229570-AAA cream.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age or older, with moderate facial acne vulgaris as defined in the protocol
* If female of childbearing potential, must take a pregnancy test and have a negative result
* Females of childbearing potential must also agree to use an adequate method of birth control, which would include:

  * systemic birth control (Subjects must have been taking the same type of birth control for at least 3 months prior to entering the study and must not change type of birth control during the study)
  * Condom with spermicide
  * IUD. Females who have had a hysterectomy, bilateral oophorectomy or bilateral tubal ligation are not required to use additional birth control methods

Exclusion Criteria:

* Known sensitivity to any of the ingredients in the study medication
* More than 3 nodulocystic acne lesions
* Use of acne treatments, therapies or medications within protocol-specified timeframes
* Presence of other skin conditions, diseases, or medical conditions that (per protocol or in the opinion of the investigator) may require concurrent therapy, interfere with the evaluation of the study medication, or compromise subject safety
* Excessive facial hair that may interfere with application of the medication and/or evaluations

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2011-03-31 (Actual); Primary Completion 2012-03-31 (Actual); Study Completion 2012-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson Varughese, Study Director — Bausch Health Americas, Inc.
Locations (18):
- United States (18):
  - University of California, San Diego, San Diego, California
  - University Clinical Trials, Inc., San Diego, California
  - Thomas J. Stephens & Associates, Inc., Colorado Springs, Colorado
  - Horizons Clinical Research Ctr., LLC, Denver, Colorado
  - North Florida Dermatology, Jacksonville, Florida
  - Hilltop Research, St. Petersburg, Florida
  - Gwinnett Clinical Research, Snellville, Georgia
  - Northwestern University, Chicago, Illinois
  - Dermatology Specialists Research, Inc, Louisville, Kentucky
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - TKL Research, Rochelle Park, New Jersey
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Wake Research Associates, Raleigh, North Carolina
  - Hilltop Research, Miamiville, Ohio
  - Penn State Medical Center, Hershey, Pennsylvania
  - Yardley Dermatology Associates, Yardley, Pennsylvania
  - Research Across America, Dallas, Texas
  - Reliance Clinical Testing Services, Irving, Texas

REFERENCES:
- See also: FDA's Drug Finder — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 investigational sites: First patient enrolled: 08 March 2011, Last patient completed: 02 March 2012
Pre-assignment Details: male and female subjects with moderate facial acne vulgaris, who met the entry criteria, were randomized with equal allocation to either 1.2%, 2.4%, or 3.6% JNJ 10229570-AAA cream or color-matched vehicle
Groups:
- 0% Facial Cream: Vehicle control Vehicle control : Color matched cream vehicle, applied once daily to the face for 12 weeks
- 1.2% Facial Cream: 1.2% JNJ 10229570-AAA 1.2% JNJ 10229570-AAA : 1.2% JNJ 10229570-AAA 1.2% cream applied once daily to the face for 12 weeks
- 2.4% Facial Cream: 2.4% JNJ 10229570-AAA 2.4% JNJ 10229570-AAA : 2.4% JNJ 10229570-AAA 2.4% cream applied once daily to the face for 12 weeks
- 3.6% Facial Cream: 3.6% JNJ 10229570-AAA 3.6% JNJ 10229570-AAA : 3.6% JNJ 10229570-AAA 3.6% cream applied once daily to the face for 12 weeks
Period: Overall Study
Arm/Group | 0% Facial Cream | 1.2% Facial Cream | 2.4% Facial Cream | 3.6% Facial Cream
Started | 106 | 109 | 109 | 107
Completed | 93 | 100 | 103 | 94
Not Completed | 13 | 9 | 6 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0% Facial Cream | 1.2% Facial Cream | 2.4% Facial Cream | 3.6% Facial Cream | Total
Number analyzed (Participants) | 106 | 109 | 109 | 107 | 431
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.9 (7.6) | 17.3 (4) | 19.7 (7) | 17.9 (5.5) | 18.7 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 45 | 51 | 53 | 198
  Male | 57 | 64 | 58 | 54 | 233
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 106 | 109 | 109 | 107 | 431

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Acne Lesion Counts
Description: Change in lesion counts between baseline and end of study
Time Frame: Baseline to Week 12
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | 0% Facial Cream | 1.2% Facial Cream | 2.4% Facial Cream | 3.6% Facial Cream
Number analyzed (Participants) | 106 | 109 | 109 | 107
Lesions | -26.0 (27.43) | -25.2 (30.23) | -29.4 (30.30) | -33.1 (29.32)

2. Secondary Outcome: Change From Baseline in the Non-inflammatory Acne Lesion Counts
Description: Change in sum of open and closed comedones.
Time Frame: Baseline through Week 12
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | 0% Facial Cream | 1.2% Facial Cream | 2.4% Facial Cream | 3.6% Facial Cream
Number analyzed (Participants) | 106 | 109 | 109 | 107
Lesions | -12.6 (20.3) | -12.0 (21.2) | -14.3 (20.9) | -15.3 (21.9)

3. Secondary Outcome: Change From Baseline in the Inflammatory Acne Lesion Counts
Description: Change in sum of papules and pustules
Time Frame: Baseline through Week 12
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | 0% Facial Cream | 1.2% Facial Cream | 2.4% Facial Cream | 3.6% Facial Cream
Number analyzed (Participants) | 106 | 109 | 109 | 107
Lesions | -13.4 (13.4) | -13.2 (16.3) | -15.1 (14.1) | -18.1 (12.9)

4. Secondary Outcome: Percent Change From Baseline in the Non-Inflammatory Acne Lesion Counts
Description: Percent Change in the Non-Inflammatory Acne Lesion Counts (the sum of open and closed comedones)
Time Frame: Baseline through Week 12
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | 0% Facial Cream | 1.2% Facial Cream | 2.4% Facial Cream | 3.6% Facial Cream
Number analyzed (Participants) | 106 | 109 | 109 | 107
Percent change | -28.6 (39.3) | -21.7 (43.1) | -31.2 (41.0) | -30.8 (37.6)

5. Secondary Outcome: Percent Change From Baseline in the Inflammatory Acne Lesion Counts
Description: Percent Change in Inflammatory Acne Lesion Counts (sum of of papules and pustules)
Time Frame: Baseline through Week 12
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | 0% Facial Cream | 1.2% Facial Cream | 2.4% Facial Cream | 3.6% Facial Cream
Number analyzed (Participants) | 106 | 109 | 109 | 107
Percent change | -39.6 (36.3) | -35.4 (45.3) | -44.7 (41.1) | -48.5 (31.9)

6. Secondary Outcome: Percent Change From Baseline in Total Acne Lesion Counts
Description: Percent change in Total Acne Lesion Counts (inflammatory lesions and non-inflammatory lesions)
Time Frame: Baseline through Week 12.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | 0% Facial Cream | 1.2% Facial Cream | 2.4% Facial Cream | 3.6% Facial Cream
Number analyzed (Participants) | 106 | 109 | 109 | 107
Percent change | -33.9 (32.7) | -27.8 (35.1) | -36.5 (36.5) | -37.7 (29.9)

ADVERSE EVENTS:
Time Frame: Through 12 weeks.
Description: Adverse events were monitored throughout the study period starting with the signing of the informed consent until completion of the last study-related procedure.
Arm/Group | 0% Facial Cream | 1.2% Facial Cream | 2.4% Facial Cream | 3.6% Facial Cream
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/109 | 0/109 | 0/107
Other Adverse Events (participants affected / at risk) | 21/106 | 17/109 | 14/109 | 15/107
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0% Facial Cream (N=106) | 1.2% Facial Cream (N=109) | 2.4% Facial Cream (N=109) | 3.6% Facial Cream (N=107)
nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 9 | 7 | 3 | 7
Headache (Nervous system disorders) | 1 | 2 | 0 | 4
Acne (Skin and subcutaneous tissue disorders) | 4 | 2 | 3 | 0
Influenza (Injury, poisoning and procedural complications) | 0 | 1 | 4 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 3
Nasal Congestion (Infections and infestations) | 2 | 3 | 0 | 0
Application Site Pruritis (General disorders) | 2 | 2 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No